CLINICAL TRIAL: NCT03634475
Title: A Safety Study of Intravitreal PP-001 in Patients With Chronic, Non-Infectious Uveitis Having Chronic Inflammation
Brief Title: A Safety Study of Intravitreal PP-001 in Patients With Chronic, Non-Infectious Uveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Panoptes Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PP-001-1001
Record Dates: First submitted 2018-08-07; First posted 2018-08-16 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-07

CONDITIONS: Non-infectious Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PP-001 (Experimental): Single intravitreal injection of 3 up to 4 doses of PP-001
  Interventions: Drug: PP-001

INTERVENTIONS:
Drug: PP-001 — Drug - no placebo

SUMMARY:
In this study, PP-001 is assessed for safety and efficacy in patients diagnosed with non-infectious chronic uveitis. PP-001 is a novel small molecule that inhibits a specific enzyme (Dihydroorotate Dehydrogenase) and has shown pre-clinical efficacy in treatment of non-infectious uveitis. PP-001 will be administered to participants as a single intravitreal injection in ascending doses.

DETAILED DESCRIPTION:
This study assesses safety and efficacy of PP-001 after intravitreal injection in patients diagnosed with non-infectious chronic uveitis. PP-001 is a novel small molecule inhibitor of Dihydroorotate Dehydrogenase (DHODH) and has shown pre-clinical efficacy in treatment of non-infectious uveitis. PP-001 is to offer a local treatment alternative to corticosteroids with the objective to reduce or possibly replace steroid intake of non-infectious uveitis patients. In the current study, PP-001 will be injected in ascending doses into the vitreous body of the eye of study participants who suffer from non-infectious uveitis. Participants will be monitored for safety and efficacy evaluation of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at the age of 18 years or older who have diagnosis of chronic, posterior uveitis, intermediate uveitis or panuveitis

Exclusion Criteria:

* Patients receiving specific medication/interventions as specified per protocol
* Pregnant or nursing patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panoptes Study Director, Study Director — Panoptes Pharma
Locations (9):
- University Hospital Vienna, Vienna, Austria
- University Hospital Leuven, Leuven, Belgium
- Germany (4):
  - Charité Berlin, Berlin
  - LMU Munich, Munich
  - University Hospital Muenster, Münster
  - University Hospital Tuebingen, Tübingen
- Rotterdam Eye Hospital, Rotterdam, Netherlands
- United Kingdom (2):
  - Bristol Eye Hospital, Bristol
  - Moorefields Eye Hospital, Moorfields

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurau S, Deuter CME, Heiligenhaus A, Pleyer U, Van Calster J, Barisani-Asenbauer T, Obermayr F, Sperl S, Seda-Zehetner R, Wildner G. A new small molecule DHODH-inhibitor [KIO-100 (PP-001)] targeting activated T cells for intraocular treatment of uveitis - A phase I clinical trial. Front Med (Lausanne). 2022 Oct 17;9:1023224. doi: 10.3389/fmed.2022.1023224. eCollection 2022. PMID 36325389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PP-001
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PP-001
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 52 [27 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety and Tolerability by Determining Treatment Emergent Adverse Events
Description: To assess safety and tolerability of ascending doses of PP-001 in participants with chronic, non-infectious uveitis when administered as single intravitreal injection
Time Frame: 40 days
Measure: Count of Participants; unit: Participants
Arm/Group | PP-001
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 14 days prior to dosing and 40 days after dosing
Arm/Group | PP-001
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PP-001 (N=12)
Conjunctival haemorrhage (Eye disorders) | 4 (5)
Anterior Chamber Cell (Eye disorders) | 3 (4)
Conjunctival hyperaemia (Eye disorders) | 3 (3)
Anterior chamber flare (Eye disorders) | 2 (2)
Eye irritation (Eye disorders) | 2 (2)
Ocular hyperaemia (Eye disorders) | 2 (2)
Punctate keratitis (Eye disorders) | 2 (3)
Conjunctival cyst (Eye disorders) | 1 (1)
Conjunctival oedema (Eye disorders) | 1 (1)
Corneal deposits (Eye disorders) | 1 (1)
Cystoid macular oedema (Eye disorders) | 1 (3)
Episcleritis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT03634475/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT03634475/SAP_001.pdf